CLINICAL TRIAL: NCT02064855
Title: The Fusion Rate With K2M VESUVIUS® Demineralized Fibers Used With K2M EVEREST® Spinal System Compared to Autologous Bone Graft With Posterior Stabilization
Brief Title: Evaluation of Fusion Rate Using K2M VESUVIUS® Demineralized Fibers With K2M EVEREST® Spinal System
Status: Terminated | Type: Observational
Why Stopped: The study was terminated early due to slow enrollment and difficulties with long-term follow-up
Sponsor: K2M, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-003
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Spinal Stenosis; Spondylolisthesis; Degenerative Disc Disease
Keywords: Spinal stenosis; Spondylolisthesis; Degenerative disc disease; Spinal fusion; Allograft; Interbody fusion
MeSH Terms: conditions — Spinal Stenosis; Spondylolisthesis; Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate fusion status and patient outcomes observed from use of the VESUVIUS Demineralized Fibers with the EVEREST Spinal System as compared to the literature reported outcomes of spinal fusion using autograft with posterior stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-cervical spinal stenosis; spondylolisthesis (grade 1 or 2); and/or degenerative disc disease (DDD) with one or two contiguous levels requiring surgical intervention between L1-S1. Qualified patients will be confirmed for inclusion by patient history and radiographic studies
* Willing and able to comply with the requirements of the protocol including follow-up requirements
* Willing and able to sign a study specific informed consent
* Skeletally mature and I 18 years old at time of enrollment

Exclusion Criteria:

* Previous spine surgery at the index level
* Previous posterior spine surgery (e.g., posterior decompression) that destabilizes the lumbar spine
* Active systemic infection or infection at the operative site
* Co-morbid medical conditions of the spine or upper/lower extremities that may affect the lumbar spine neurological and/or pain assessment
* Metabolic bone disease such as osteoporosis and osteopenia that contradicts spinal surgery
* History of an osteoporotic fracture
* History of an endocrine or metabolic disorder (e.g., Paget's disease) known to affect bone and mineral metabolism
* Taking medications that may interfere with bony/soft tissue healing including chronic steroid use
* Known allergy to titanium or cobalt chrome
* Rheumatoid arthritis or other autoimmune disease or a systemic disorder such as HIV, active hepatitis B or C, or fibromyalgia
* Insulin-dependent type 1 or type 2 diabetes
* Medical condition (e.g., unstable cardiac disease, cancer) that may result in patient death or have an effect on outcomes prior to study completion
* Pregnant, or intends to become pregnant, during the course of the study
* Severe obesity (Body Mass Index > 40)
* Physical or mental condition (e.g., psychiatric disorder, senile dementia, Alzheimer's disease, alcohol or drug addiction) that would interfere with patient self-assessment of function, pain, or quality of life.
* Involved in current or pending spinal litigation where permanent disability benefits are being sought
* Incarcerated at the time of study enrollment
* Current participation in an investigational study that may impact study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified from the surgeon's practice.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-12-12 (Actual)

REFERENCES:
- [Background] Cammisa FP Jr, Lowery G, Garfin SR, Geisler FH, Klara PM, McGuire RA, Sassard WR, Stubbs H, Block JE. Two-year fusion rate equivalency between Grafton DBM gel and autograft in posterolateral spine fusion: a prospective controlled trial employing a side-by-side comparison in the same patient. Spine (Phila Pa 1976). 2004 Mar 15;29(6):660-6. doi: 10.1097/01.brs.0000116588.17129.b9. PMID 15014276
- [Background] Chen WJ, Tsai TT, Chen LH, Niu CC, Lai PL, Fu TS, McCarthy K. The fusion rate of calcium sulfate with local autograft bone compared with autologous iliac bone graft for instrumented short-segment spinal fusion. Spine (Phila Pa 1976). 2005 Oct 15;30(20):2293-7. doi: 10.1097/01.brs.0000182087.35335.05. PMID 16227892
- [Background] Glassman SD, Dimar JR, Carreon LY, Campbell MJ, Puno RM, Johnson JR. Initial fusion rates with recombinant human bone morphogenetic protein-2/compression resistant matrix and a hydroxyapatite and tricalcium phosphate/collagen carrier in posterolateral spinal fusion. Spine (Phila Pa 1976). 2005 Aug 1;30(15):1694-8. doi: 10.1097/01.brs.0000172157.39513.80. PMID 16094268
- [Background] Vaccaro AR, Anderson DG, Patel T, Fischgrund J, Truumees E, Herkowitz HN, Phillips F, Hilibrand A, Albert TJ, Wetzel T, McCulloch JA. Comparison of OP-1 Putty (rhBMP-7) to iliac crest autograft for posterolateral lumbar arthrodesis: a minimum 2-year follow-up pilot study. Spine (Phila Pa 1976). 2005 Dec 15;30(24):2709-16. doi: 10.1097/01.brs.0000190812.08447.ba. PMID 16371892
- [Background] Dimar JR, Glassman SD, Burkus KJ, Carreon LY. Clinical outcomes and fusion success at 2 years of single-level instrumented posterolateral fusions with recombinant human bone morphogenetic protein-2/compression resistant matrix versus iliac crest bone graft. Spine (Phila Pa 1976). 2006 Oct 15;31(22):2534-9; discussion 2540. doi: 10.1097/01.brs.0000240715.78657.81. PMID 17047540
- [Background] Niu CC, Tsai TT, Fu TS, Lai PL, Chen LH, Chen WJ. A comparison of posterolateral lumbar fusion comparing autograft, autogenous laminectomy bone with bone marrow aspirate, and calcium sulphate with bone marrow aspirate: a prospective randomized study. Spine (Phila Pa 1976). 2009 Dec 1;34(25):2715-9. doi: 10.1097/BRS.0b013e3181b47232. PMID 19940728
- [Background] Taghavi CE, Lee KB, Keorochana G, Tzeng ST, Yoo JH, Wang JC. Bone morphogenetic protein-2 and bone marrow aspirate with allograft as alternatives to autograft in instrumented revision posterolateral lumbar spinal fusion: a minimum two-year follow-up study. Spine (Phila Pa 1976). 2010 May 15;35(11):1144-50. doi: 10.1097/BRS.0b013e3181bb5203. PMID 20139805

RESULTS

PARTICIPANT FLOW:
Groups:
- EVEREST/VESUVIUS Demineralized Fibers: This group involves patients treated with the VESUVIUS Demineralized Fibers and EVEREST system that had:
  1. Diagnosis of spinal stenosis, spondylolisthesis (grade 1 or 2), and/or degenerative disc disease (DDD).
  2. Qualified for inclusion by patient history and radiographic studies.
  3. One or two contiguous levels requiring surgical intervention between L1-S1 Skeletally mature and greater than or equal to 18 years old at time of enrollment
Period: Overall Study
Arm/Group | EVEREST/VESUVIUS Demineralized Fibers
Started | 108
Completed | 53
Not Completed | 55

BASELINE CHARACTERISTICS:
Groups:
- Demographics and Baseline Characteristics: Demographics and Baseline Characteristics (Patient Population)
Arm/Group | Demographics and Baseline Characteristics
Number analyzed (Participants) | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 63
  >=65 years | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.45 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 52
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The study Case Report Forms did not include Race/Ethnicity
Region of Enrollment [Number; unit: participants]
  United States | 108
Height [Mean (Standard Deviation); unit: inches] | 66.57 (4.09)
Weight [Mean (Standard Deviation); unit: pounds] | 187.19 (37.67)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: lbs/(in^2)*703] | 29.61 (4.86)
Tobacco Use [Count of Participants; unit: Participants]
  Never | 47
  Quit | 45
  Currently Use | 16
  Missing | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: All adverse events will be documented including device related, procedure related and additional serious adverse events.
Time Frame: 24 months
Measure: Number; unit: participants
Groups:
- Up to Post Operative: AEs and SAEs that occurred at the beginning of the study up to Post Operative
- Post-Operative to 3 Months: AEs and SAEs that occurred at the beginning of the study from Post-Operative to 3 Months
- 3 to 6 Months: AEs and SAEs that occurred at the beginning of the study from 3 to 6 Months
- 6 to 12 Months: AEs and SAEs that occurred at the beginning of the study from 6 to 12 Months
- 12 to 24+ Months: AEs and SAEs that occurred at the beginning of the study from 12 to 24+ Months
- Overall: Overall AEs and SAEs
Arm/Group | Up to Post Operative | Post-Operative to 3 Months | 3 to 6 Months | 6 to 12 Months | 12 to 24+ Months | Overall
Number analyzed (Participants) | 108 | 108 | 108 | 108 | 108 | 108
participants
  Any AE | 51 | 15 | 19 | 23 | 24 | 76
  Any AE: Procedure Related | 28 | 0 | 1 | 1 | 4 | 50
  Any AE: Device Related | 2 | 0 | 0 | 0 | 1 | 3
  Any AE: Mild | 21 | 5 | 4 | 5 | 8 | 36
  Any AE: Moderate | 34 | 10 | 14 | 17 | 17 | 60
  Any AE: Severe | 10 | 0 | 4 | 4 | 2 | 19
  Any SAE | 16 | 0 | 4 | 5 | 3 | 25
  Any SAE: Procedure Related | 10 | 0 | 0 | 0 | 1 | 11
  Any SAE: Device Related | 2 | 0 | 0 | 0 | 0 | 2
  Any SAE: Mild | 3 | 0 | 0 | 0 | 0 | 3
  Any SAE: Moderate | 6 | 0 | 2 | 2 | 1 | 11
  Any SAE: Severe | 7 | 0 | 1 | 3 | 2 | 12

2. Primary Outcome: Fusion Status on CT at 12 Months
Description: Fusion is categorized as Partial consolidation and Bridging/Fusion. Partial consolidation is defined as consolidation of bone graft material with no complete bridging seen. Bridging/Fusion is defined as clear evidence of solid bridging bone between posterolateral gutters, facet joints and/or transverse processes.
Time Frame: 12 months
Population: Image Assessed at Visit
Measure: Count of Units; unit: Number of Image Assessed
Units Other Than Participants: Number of Image Assessed
Groups:
- Fusion Assessment: Fusion status of participants on CT assessed at 12 month visit
Arm/Group | Fusion Assessment
Number analyzed (Participants) | 108
Number analyzed (Number of Image Assessed) | 80
Number of Image Assessed
  Fused | 63
  Not Fused | 17

3. Secondary Outcome: Radiographic Assessments
Description: X-rays at pre-operative and post operative include: AP& Lateral; Flex/Ext & Oblique X-rays. Radiographic assessments being performed include:
  * Posterior/Transverse process fusion, Right side (by level)
  * Posterior/Transverse process fusion, Left side (by level)
  * Anterior fusion, if TLIF procedure done, by level
  * Overall fusion by level
  * Device Condition
  * Device Subsidence
  * Device Migration
Time Frame: 12m
Population: Each Arm/group has different overall number of participants assessed.
Measure: Count of Participants; unit: Participants
Groups:
- Graft Ratio; Instrumented Levels; Vertebrae Levels: Radiographic Assessment of the fusion at 12 months
Arm/Group | Graft Ratio | Instrumented Levels | Vertebrae Levels
Number analyzed (Participants) | 84 | 84 | 104
Participants
  3:2 (Vesuvius Fibers: BMA): number analyzed (Participants) | 31 | 0 | 0
  3:2 (Vesuvius Fibers: BMA): Bridging/Fusion | 13 |  |
  3:2 (Vesuvius Fibers: BMA): Partial Consolidation | 13 |  |
  3:2 (Vesuvius Fibers: BMA): Absent | 4 |  |
  3:2 (Vesuvius Fibers: BMA): Unknown | 1 |  |
  1:1 (Vesuvius Fibers: BMA): number analyzed (Participants) | 26 | 0 | 0
  1:1 (Vesuvius Fibers: BMA): Bridging/Fusion | 7 |  |
  1:1 (Vesuvius Fibers: BMA): Partial Consolidation | 9 |  |
  1:1 (Vesuvius Fibers: BMA): Absent | 9 |  |
  1:1 (Vesuvius Fibers: BMA): Unknown | 1 |  |
  Other: number analyzed (Participants) | 27 | 0 | 0
  Other: Bridging/Fusion | 11 |  |
  Other: Partial Consolidation | 9 |  |
  Other: Absent | 5 |  |
  Other: Unknown | 2 |  |
  1 Level: number analyzed (Participants) | 0 | 64 | 0
  1 Level: Bridging/Fusion |  | 27 |
  1 Level: Partial Consolidation |  | 21 |
  1 Level: Absent |  | 13 |
  1 Level: Unknown |  | 3 |
  2 Levels: number analyzed (Participants) | 0 | 20 | 0
  2 Levels: Bridging/Fusion |  | 3 |
  2 Levels: Partial Consolidation |  | 12 |
  2 Levels: Absent |  | 4 |
  2 Levels: Unknown |  | 1 |
  L3-L4: number analyzed (Participants) | 0 | 0 | 14
  L3-L4: Bridging/Fusion |  |  | 5
  L3-L4: Partial Consolidation |  |  | 7
  L3-L4: Absent |  |  | 2
  L3-L4: Unknown |  |  | 0
  L4-L5: number analyzed (Participants) | 0 | 0 | 63
  L4-L5: Bridging/Fusion |  |  | 22
  L4-L5: Partial Consolidation |  |  | 25
  L4-L5: Absent |  |  | 12
  L4-L5: Unknown |  |  | 4
  L5-S1: number analyzed (Participants) | 0 | 0 | 27
  L5-S1: Bridging/Fusion |  |  | 7
  L5-S1: Partial Consolidation |  |  | 11
  L5-S1: Absent |  |  | 8
  L5-S1: Unknown |  |  | 1

4. Secondary Outcome: Radiographic Assessments
Description: X-rays at post operative include: AP& Lateral; Flex/Ext & Oblique X-rays. Radiographic assessments being performed include:
  Device Condition Device Subsidence Device Migration
Time Frame: 12 Months and 24 Months
Population: The participants data analyzed differ from the overall number of participants for the Arms. Cages were optional per protocol as such the decrease in the number of participants.
Measure: Count of Participants; unit: Participants
Groups:
- Level 1; Level 2: Superior; Level 2: Inferior: Radiographic assessments performed to determine Device Condition
Arm/Group | Level 1 | Level 2: Superior | Level 2: Inferior
Number analyzed (Participants) | 79 | 29 | 29
Participants
  12 Mo Hardware Condition: number analyzed (Participants) | 64 | 21 | 21
  12 Mo Hardware Condition: Intact | 51 | 16 | 19
  12 Mo Hardware Condition: Loosening | 12 | 4 | 1
  12 Mo Hardware Condition: Fracture | 1 | 0 | 0
  12 Mo Hardware Condition: Absent | 0 | 0 | 0
  12 Mo Hardware Condition: Partial Consolidation | 0 | 0 | 0
  12 Mo Hardware Condition: Bridging/Fusion | 0 | 0 | 0
  12 Mo Hardware Condition: Unable to assess | 0 | 1 | 1
  24 Mo Hardware Condition: number analyzed (Participants) | 39 | 14 | 14
  24 Mo Hardware Condition: Intact | 32 | 10 | 13
  24 Mo Hardware Condition: Loosening | 4 | 4 | 1
  24 Mo Hardware Condition: Fracture | 1 | 0 | 0
  24 Mo Hardware Condition: Absent | 0 | 0 | 0
  24 Mo Hardware Condition: Partial Consolidation | 0 | 0 | 0
  24 Mo Hardware Condition: Bridging/Fusion | 0 | 0 | 0
  24 Mo Hardware Condition: Unable to assess | 2 | 0 | 0
  12 Mo Cage Condition: number analyzed (Participants) | 22 | 10 | 12
  12 Mo Cage Condition: Intact | 0 | 0 | 0
  12 Mo Cage Condition: Loosening | 0 | 0 | 0
  12 Mo Cage Condition: Fracture | 0 | 0 | 0
  12 Mo Cage Condition: Absent | 8 | 2 | 4
  12 Mo Cage Condition: Partial Consolidation | 3 | 5 | 4
  12 Mo Cage Condition: Bridging/Fusion | 10 | 2 | 3
  12 Mo Cage Condition: Unable to assess | 1 | 1 | 1
  24 Mo Cage Condition: number analyzed (Participants) | 17 | 6 | 7
  24 Mo Cage Condition: Intact | 0 | 0 | 0
  24 Mo Cage Condition: Loosening | 0 | 0 | 0
  24 Mo Cage Condition: Fracture | 0 | 0 | 0
  24 Mo Cage Condition: Absent | 3 | 1 | 1
  24 Mo Cage Condition: Partial Consolidation | 1 | 2 | 2
  24 Mo Cage Condition: Bridging/Fusion | 12 | 2 | 3
  24 Mo Cage Condition: Unable to assess | 1 | 1 | 1

5. Secondary Outcome: Change From Baseline in Daily Functional Ability Scores on the Oswestry Disability Index (ODI)
Description: This patient-reported outcome measure is a 10 item questionnaire that evaluates disability and functional impairment associated with back problems. Each item is scored from 0 up to 5, with higher scores corresponding to greater disability. A total ODI score is determined by adding the scores of the individual questions and dividing that total by the maximum possible score (i.e., 50 if all questions are answered) to yield a percentage. Therefore, the ODI score ranges from 0% to 100%.
Time Frame: Baseline (Pre-Op), 24 months
Population: While 53 participants completed the study, 1 patient did not complete the survey at 24 Month.
  2 patient did not complete the survey at 12 Month. 5 patient did not complete the survey at 6 Month. 4 patient did not complete the survey at 3 Month. 2 patient did not complete the survey at Initial Post-Op.
  1 patient did not complete the survey at Pre-Op.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-Operative: Daily Functional Ability Scores on the Oswestry Disability Index (ODI)
- Initial Post Operative; 3 Month; 6 Month; 12 Month; 24 Month: Change From Baseline in Daily Functional Ability Scores on the Oswestry Disability Index (ODI)
Arm/Group | Pre-Operative | Initial Post Operative | 3 Month | 6 Month | 12 Month | 24 Month
Number analyzed (Participants) | 107 | 101 | 98 | 90 | 83 | 52
score on a scale
  Baseline | 45.1 (17.2) | 36.4 (19.5) | 24.3 (18.3) | 20.5 (18.2) | 18.0 (18.3) | 16.6 (18.4)
  Change from Baseline | NA (NA) — This field is not applicable as it is the baseline and there would not be any change from the baseline | -8.0 (20.9) | -20.3 (19.9) | -24.4 (19.7) | -25.8 (18.9) | -26.3 (21.0)

6. Secondary Outcome: Change From Baseline in Pain Scores on the Visual Analog Scale (VAS) at 24 Months
Description: VAS scale ranged from 0 to 100mm with the 100mm accounting for the highest level of pain
Time Frame: Baseline (up to 8 weeks post-operatively) to 24 months
Population: While 53 participants completed the study, 1-2 patients did not complete the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Back; Left Hip; Right Hip; Left Leg; Right Leg: Change from baseline in pain scores on the Visual Analog Scale (VAS) at 24 months
Arm/Group | Back | Left Hip | Right Hip | Left Leg | Right Leg
Number analyzed (Participants) | 52 | 51 | 52 | 51 | 51
score on a scale | -44.3 (30.51) | -38.6 (35.82) | -27.9 (39.02) | -37.9 (38.90) | -36.1 (42.90)

7. Secondary Outcome: Change From Baseline in Quality of Life Scores on the SF-12v2 at 24 Months
Description: SF-12v2 ranged between 0 and 100 points. The higher the points the better the self-assessed quality of life.
Time Frame: Baseline (up to 8 weeks post-operatively) to 24 months
Population: While 53 participants completed the study, 1 patient did not complete the survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mental Health; Physical Health: Change From Baseline in Quality of Life Scores on the SF-12v2 at 24 Months
Arm/Group | Mental Health | Physical Health
Number analyzed (Participants) | 52 | 52
score on a scale | 4.603 (10.257) | 11.734 (10.042)

8. Secondary Outcome: Patient Satisfaction
Description: Patient Satisfaction at 12 Mo and 24 Mo
Time Frame: 12 months, 24 months
Population: All participants for both intervals filled out the surveys
Measure: Count of Participants; unit: Participants
Groups:
- 12 Month: Patient Satisfaction at 12 Mo
- 24 Month: Patient Satisfaction at 24 Mo
Arm/Group | 12 Month | 24 Month
Number analyzed (Participants) | 85 | 53
Participants
  Satisfied: Yes | 72 | 43
  Satisfied: No | 5 | 6
  Satisfied: Not Reported | 8 | 4
  Repeat Procedure: Yes | 71 | 45
  Repeat Procedure: No | 5 | 4
  Repeat Procedure: Not Reported | 9 | 4

9. Secondary Outcome: Length of Surgery Time
Description: The length of the surgical procedure from the initial incision to final closure.
Time Frame: At time of surgery
Population: 5 Subjects did not have a surgical time recorded
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Surgery Time: Length of Surgery Time
Arm/Group | Surgery Time
Number analyzed (Participants) | 103
Hours | 3.12 (1.29)

10. Secondary Outcome: Length of Anesthesia Time
Description: The length of time the patient is under anesthesia.
Time Frame: At time of surgery
Population: 6 Subjects did not have anesthesia time recorded
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Anesthesia Time: Length of Anesthesia Time
Arm/Group | Anesthesia Time
Number analyzed (Participants) | 102
Hours | 4.23 (1.40)

11. Secondary Outcome: Estimated Blood Loss
Description: The amount of blood loss over the entire length of the surgery
Time Frame: At time of surgery
Population: 1 Subject did not have the amount of blood loss recorded
Measure: Mean (Standard Deviation); unit: Cubic Centimeters
Groups:
- Estimated Blood Loss: The amount of blood loss over the entire length of the surgery will be captured.
Arm/Group | Estimated Blood Loss
Number analyzed (Participants) | 107
Cubic Centimeters | 250.50 (238.79)

12. Secondary Outcome: Length of Hospital Stay
Description: The length of the hospital stay from the date of admission to the date of discharge .
Time Frame: Admission to discharge
Population: All patients are accounted for
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Length of Hospital Stay: The length of Hospital Stay
Arm/Group | Length of Hospital Stay
Number analyzed (Participants) | 108
Days | 4.15 (1.83)

13. Secondary Outcome: Time to Return to Work/School
Description: The ability to and the time it takes for the subject to be cleared to return to work/school from the date of surgery by looking at the percentage increase of participants who were able to return to work without any restrictions.
Time Frame: Pre-Op to 24 months
Population: Includes all participants who returned for each visit interval with those who did not respond to this question accounted for in the missing row.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Operative; Initial Post Operative; 3 Month; 6 Month; 12 Month; 24 Month: Time to Return to Work/School
Arm/Group | Pre-Operative | Initial Post Operative | 3 Month | 6 Month | 12 Month | 24 Month
Number analyzed (Participants) | 108 | 103 | 100 | 95 | 85 | 53
Participants
  Unemployment, unrelated to back/leg conditions | 21 | 19 | 20 | 23 | 15 | 2
  Not attending work/school by choice | 22 | 24 | 22 | 19 | 17 | 16
  Unable to go due to back/leg pain/conditions | 14 | 43 | 15 | 3 | 4 | 5
  Attending work/school with some restrictions | 20 | 15 | 24 | 18 | 10 | 1
  Attending work/school with no restrictions | 31 | 2 | 19 | 28 | 36 | 28
  Missing | 0 | 0 | 0 | 4 | 3 | 1

14. Secondary Outcome: Use of Narcotics Post-surgery
Description: The types and dosages of any narcotics taken by the patient post-surgery will be documented.
Time Frame: Pre-Op to 24 months
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Groups:
- Pre-Operative; Initial Post Operative; 3 Month; 6 Month; 12 Month; 24 Month: Use of Narcotics Post-surgery
Arm/Group | Pre-Operative | Initial Post Operative | 3 Month | 6 Month | 12 Month | 24 Month
Number analyzed (Participants) | 108 | 103 | 100 | 95 | 85 | 53
Participants
  Back Meds: None | 11 | 9 | 24 | 34 | 43 | 27
  Back Meds: Non-narcotics or NSAIDs | 42 | 15 | 32 | 32 | 23 | 19
  Back Meds: Intermittent short-acting narcotics | 20 | 37 | 23 | 14 | 7 | 2
  Back Meds: Chronic daily short-acting narcotics | 26 | 36 | 16 | 12 | 7 | 2
  Back Meds: Chronic daily long-acting narcotics | 5 | 6 | 5 | 1 | 3 | 1
  Back Meds: IV or injected narcotics | 1 | 0 | 0 | 0 | 0 | 0
  Back Meds: Epidural/Facet injections | 3 | 0 | 0 | 0 | 1 | 0
  Back Meds: Missing | 0 | 0 | 0 | 2 | 1 | 2
  Non-Back Meds: None | 79 | 80 | 81 | 64 | 60 | 36
  Non-Back Meds: Non-narcotics or NSAIDs | 20 | 15 | 14 | 25 | 16 | 14
  Non-Back Meds: Intermittent short-acting narcotics | 6 | 7 | 2 | 4 | 5 | 0
  Non-Back Meds: Chronic daily short-acting narcotics | 2 | 0 | 2 | 0 | 3 | 1
  Non-Back Meds: Chronic daily long-acting narcotics | 1 | 1 | 1 | 0 | 0 | 0
  Non-Back Meds: IV or injected narcotics | 0 | 0 | 0 | 0 | 0 | 0
  Non-Back Meds: Epidural/Facet injections | 0 | 0 | 0 | 0 | 0 | 0
  Non-Back Meds: Missing | 0 | 0 | 0 | 2 | 1 | 2

ADVERSE EVENTS:
Time Frame: From Operative to 24+ Months
Description: Any untoward medical occurrence in a subject undergoing surgery in this trial which does not necessarily have a causal relationship with this intervention. An AE can, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the one of the devices. Any AE that occurs during the subject's participation in the study will be recorded on the Adverse Event case report form.
Groups:
- Participants With Adverse Events: Participants were evaluated for all adverse events including device related, procedure related, and additional serious adverse events.
  3 of the 25 SAE participants did not experience a non-SAE events. The other 22 participants had events in both categories.
  The study did not establish a frequency threshold, therefore, all AEs are listed.
Arm/Group | Participants With Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/108
Serious Adverse Events (participants affected / at risk) | 25/108
Other Adverse Events (participants affected / at risk) | 73/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adverse Events (N=108)
Coronary artery disease (Cardiac disorders) | 1 (1)
Gastrointestinal anastomotic stenosis (Gastrointestinal disorders) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lung Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cervical radiculopathy (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Gallbladder disorder (Hepatobiliary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Post procedural (Injury, poisoning and procedural complications) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1)
Kyphosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Dural tear (Nervous system disorders) | 1 (1)
Device failure (Product Issues) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Iliac vein perforation (Vascular disorders) | 1 (1)
Myocardial infarction (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With Adverse Events (N=108)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Eye contusion (Eye disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Functional gastrointestinal disorder (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Chest Pain (General disorders) | 3 (3)
Fatigue (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Impaired healing (General disorders) | 4 (5)
Incision site impaired healing (General disorders) | 1 (2)
Pain (General disorders) | 1 (2)
Peripheral swelling (General disorders) | 4 (5)
Post procedural fever (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 6 (9)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Implant site erosion (Injury, poisoning and procedural complications) | 1 (1)
incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Rotator cuff syndrome (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 2 (2)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Body temperature increased (Investigations) | 1 (2)
Culture negative (Investigations) | 1 (1)
Electrocardiogram (Investigations) | 1 (1)
Electrocardiogram ambulatory (Investigations) | 1 (1)
Lasegue's test positive (Investigations) | 2 (3)
Diabetic neuropathy (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17)
Back Pain (Musculoskeletal and connective tissue disorders) | 27 (33)
Coccydynia (Musculoskeletal and connective tissue disorders) | 4 (4)
Gout (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Incomplete spinal fusion (Musculoskeletal and connective tissue disorders) | 2 (3)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb asymmetry (Musculoskeletal and connective tissue disorders) | 1 (1)
Lower limb fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle strain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (5)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 (10)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19 (24)
Restless legs syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Sacroilitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Sciatica (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Wrist fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 (2)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Dural tear (Nervous system disorders) | 4 (4)
Dysaesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
hypoaesthesia (Nervous system disorders) | 6 (6)
Lumbar radiculopathy (Nervous system disorders) | 2 (2)
Lumbar spinal stenosis (Nervous system disorders) | 3 (3)
Nerve compression (Nervous system disorders) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3)
Incision site impaired healing (Injury, poisoning and procedural complications) | 1 (1)
Confusion postoperative (Psychiatric disorders) | 1 (1)
Bladder dysfunction (Renal and urinary disorders) | 1 (1)
Calculus urinal (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Nervous system disorders) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (1)
Testicular swelling (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Basal cell carcinoma (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (4)
Skin laceration (Skin and subcutaneous tissue disorders) | 1 (1)
Incisional drainage (Surgical and medical procedures) | 1 (2)
Contusion (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 1 (1)
Perthes disease (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution/PI shall not disclose/use any confidential/proprietary information (CI) disclosed to/developed by the Institution during the study. Institution/PI agree to hold the results of the Study in confidence, and shall not disclose them except with prior written consent of K2M. Institution agrees to submit any Articles to K2M for review prior to publication and agrees to edit out any confidential information identified by K2M.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT02064855/Prot_SAP_000.pdf